CLINICAL TRIAL: NCT05219071
Title: Transdermal Rigidity Assessment Via Ischemia (and Temperature) of the Penis (TRIP) Versus the Rigiscan: A New Sensor-driven Device to Measure Rigidity of the Penis
Brief Title: TRIP-Patch vs the Rigiscan
Acronym: TRIP-Patch
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Evelien Trip, Principal Investigator, St. Antonius Hospital
Other Study IDs: 75891
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Erectile Dysfunction
Keywords: Rigiscan; Nocturnal erection; Temperature; Saturation
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In men without erectile problems, night time erections occur during the REM-sleep. For this study the current diagnostic test, the Rigiscan is compared, with the data from the TRIP-Patch during the night. To validate discriminating sensor-readings between flaccid state and full rigidity of the penis. Eventually, to have a validated device, a patch in the size of a postage stamp, that easily measures erectile function at home. Furthermore the temperature on the outside of the thigh will be measured.

DETAILED DESCRIPTION:
Background of the study: Erectile dysfunction (ED) is defined as the persistent or recurrent inability to attain and maintain an erection sufficient to perform sexual activity. ED has an effect on physical and psychosocial well-being. The current diagnostic test, the Rigiscan to measure night time erections, has a lot of disadvantages.

When an erection occurs and there is no inflow and outflow in the corpora cavernosa it is expected that the saturation will drop. As known with low flow priapism. From a study from Solnick, the mean skin temperature in younger male (19-33 years old) increases from 33,8°C to 36.2°C during arousal. A penile oximeter and temperature sensor was developed, to measure saturation and temperature of the penis during the night. The TRIP-Patch (Transdermal Rigidity assessment via Ischemia of the Penis) is expected to continuously measure saturation levels in the corpora cavernosa by real time monitoring with a photodiodes and LEDs and the sensor has a temperature logger.

Objective of the study: see above Study design: Observational study Study population: Healthy volunteers are asked to participate after informed consent. Age between 18 and 40 years. Both sensors and the Rigiscan will be placed at the same time, when 10 patients have night time erections with the Rigiscan, the study is complete.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without (a history of) erectile dysfunction
* Signed informed consent
* Male
* Between 18-40 year

Exclusion Criteria:

* Volunteers who are unwilling to sign written informed consent
* Volunteers with sickle cell anemia because this could affect the accuracy of the measurements
* Volunteers with erectile dysfunction

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents and medical students in the St Antonius Hospital and other volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Change in saturation | 1 night
  Change in saturation of corpora cavernosa during an erection
temperature change | 1 night
  Change in penile skin temperature during an erection

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Trip, drs, MD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No